CLINICAL TRIAL: NCT03374631
Title: Stimulating the Social Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Amy Pinkham, PhD, Associate Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-126
Record Dates: First submitted 2017-12-07; First posted 2017-12-15 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Healthy Adults

STUDY DESIGN:
Intervention Model Description: Participants will complete active and sham simulation sessions in a randomized, counterbalanced order approximately one week apart.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active anodal tDCS, Then Sham tDCS (Experimental): Active anodal tDCS followed by behavioral testing; one week later, sham tDCS followed by behavioral testing
  Interventions: Device: active anodal tDCS; Device: sham tDCS
- Sham tDCS, then Active anodal tDCS (Sham Comparator): Sham tDCS followed by behavioral testing; one week later, active anodal tDCS followed by behavioral testing.
  Interventions: Device: active anodal tDCS; Device: sham tDCS

INTERVENTIONS:
Device: active anodal tDCS — active anodal tDCS with behavioral tasks and self-report measures to assess paranoid ideation
Device: sham tDCS — sham tDCS with behavioral tasks and self-report measures to assess paranoid ideation

SUMMARY:
This study investigates whether the way in which individuals process social stimuli can be altered, and specifically, whether feelings of paranoia and suspiciousness can be reduced by stimulating the brain's regulatory regions via transcranial Direct Current Stimulation (tDCS).

DETAILED DESCRIPTION:
Although paranoid ideation is typically associated with severe mental illnesses such as schizophrenia or bipolar disorder, 10-15% of individuals in the general population report experiencing paranoid thoughts on a regular basis. These individuals who are high in sub-clinical paranoia can show impaired work and social functioning as compared to individuals low in sub-clinical paranoia. The wide spread prevalence and negative functional impact of heightened paranoia reinforces the need to develop interventions that may help to reduce problematic patterns of paranoid thinking in both healthy individuals and those with mental illness.

Transcranial Direct Current Stimulation (tDCS) is a form of noninvasive neurostimulation which has been proposed as a therapeutic procedure in numerous psychiatric conditions. TDCS therefore may be a promising therapeutic technique for reducing symptoms of psychosis, and specifically paranoia. This study will compare experiences of paranoid ideation in individuals who are high in sub-clinical paranoia across two conditions: active anodal tDCS and sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 ad 35
* previous classification as being high in sub-clinical paranoia

Exclusion Criteria:

* diagnosis of mental illness
* use of psychotropic medication
* Presence or history of medical, cardiac, or neurological disorders that may affect brain function (e.g., cardiac disease, endocrine disorders, renal disease, pulmonary disease, history of seizures or head trauma with unconsciousness for a period of 15 minutes or greater or CNS tumors)
* Presence of sensory limitation including visual (e.g., blindness, glaucoma, vision uncorrectable to 20/40) or hearing (e.g. hearing loss) impairments that interfere with assessment
* Not proficient in English
* Contraindications for tDCS (e.g., pregnancy or implanted devices such as pace maker)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Pinkham, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The Unversity of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (20 Minutes)
Arm/Group | Active Anodal tDCS, Then Sham tDCS | Sham tDCS, Then Active Anodal tDCS
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Active Anodal tDCS, Then Sham tDCS | Sham tDCS, Then Active Anodal tDCS
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Intervention (20 Minutes)
Arm/Group | Active Anodal tDCS, Then Sham tDCS | Sham tDCS, Then Active Anodal tDCS
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Anodal tDCS, Then Sham tDCS | Sham tDCS, Then Active Anodal tDCS | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (2.30) | 19.6 (1.98) | 20.15 (2.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 10 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 7 | 13
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in General Paranoid Ideation for Active vs. Sham Simulation
Description: Level of paranoid ideation will be assessed with the self-report Paranoia Scale (PS; Fenigstein & Vanable, 1992) both before and after tDCS to assess changes related to tDCS. The PS is a self-report measure designed to assess sub-clinical paranoid thought. Scores range from 20-100 with higher scores indicating higher levels of paranoia. The amount of pre-post change (i.e. PS score assessed before stimulation minus score after stimulation) is the primary value of interest and will be compared between active and sham stimulation. Improvements in paranoia will be indicated by positive values.
Time Frame: Paranoid ideation will be assessed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Stimulation: 20 minutes of Active anodal tDCS followed by behavioral testing
- Sham Stimulation: 20 minutes of Sham tDCS followed by behavioral testing
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 40 | 40
score on a scale | 1.60 (3.11) | .73 (3.80)

2. Primary Outcome: Change in Change in Social Paranoia for Active vs. Sham Simulation
Description: Level of paranoid ideation will be assessed with the persecution subscale of the State Social Paranoia Scale (SSPS: Freeman et al., 2007) both before and after tDCS to assess changes related to tDCS. The SSPS is a psychometrically sound 20-item self- report measure assessing current levels of paranoid, positive, and neutral thinking about others. Ten items comprise the persecution subscale, and scores on this subscale range from 10-50 with higher scores indicating greater paranoia. The amount of pre-post change (i.e.SSPS score before stimulation minus SSPS score after stimulation) will be compared between active and sham stimulation. Positive values indicate reductions in paranoia after stimulation.
Time Frame: Paranoid ideation will be assessed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Anodal Stimulation: 20 minutes of Active anodal tDCS followed by behavioral testing
- Sham tDCS: 20 minutes of Sham tDCS followed by behavioral testing
Arm/Group | Active Anodal Stimulation | Sham tDCS
Number analyzed (Participants) | 40 | 40
score on a scale | .75 (2.52) | .93 (2.34)

3. Secondary Outcome: Trustworthiness Task Score for Active vs. Sham Stimulation
Description: Participants will complete the Trustworthiness Task (Adolphs, Tranel, & Damasio, 1998), which asks individuals to view 42 images of others and rate their level of trustworthiness on a scale from -3 to 3. Scores range from -126 to 126. Higher scores indicate greater perceptions of trustworthiness. Mean ratings following each stimulation type (active vs. sham) are calculated.
Time Frame: assessed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Anodal tDCS: 20 minutes of Active anodal tDCS followed by behavioral testing
Arm/Group | Active Anodal tDCS | Sham tDCS
Number analyzed (Participants) | 40 | 40
score on a scale | -.14 (.64) | -.14 (.60)

4. Secondary Outcome: Penn Emotion Recognition Test for Active vs. Sham Stimulation
Description: The Emotion Recognition 40 (ER-40; Kohler, Turner, Bilker, Brinsinger, Siegel, Kanes... Gur, 2003) is a standardized, computer administered measure of facial affect recognition ability. It includes 40 color photographs of faces expressing 4 basic emotions (i.e. happiness, sadness, anger or fear) and neutral expressions. Participants view one face at a time and are asked to choose the correct emotion for each face. Scores range from 0-40 with higher scores indicating better accuracy. Mean performance following each stimulation type (active vs. sham) are calculated.
Time Frame: assessed 30 minutes after completion of the active/sham stimulation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Anodal tDCS | Sham tDCS
Number analyzed (Participants) | 40 | 40
score on a scale | 35.05 (2.39) | 35.33 (2.31)

ADVERSE EVENTS:
Time Frame: 10 days for each arm.
Arm/Group | Active Anodal tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT03374631/Prot_SAP_000.pdf